CLINICAL TRIAL: NCT07100548
Title: Mental Health in the Digital Age: A Qualitative Study of Youth Responses to Depression Education Delivered on Social Media
Brief Title: A Qualitative Analysis of Youth Responses to Depression Education Delivered on Social Media
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Prof. Otto Beisheim Foundation (Other)
Responsible Party: Principal Investigator, Ellen Greimel, Working group leader, Ludwig-Maximilians - University of Munich
Other Study IDs: 25-0088
Record Dates: First submitted 2025-07-24; First posted 2025-08-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Depressive Disorder; Depression - Major Depressive Disorder; Depression in Adolescence
Keywords: depression; prevention; social media; adolescents; depression literacy; stigma; help-seeking; psychoeducation
MeSH Terms: conditions — Depressive Disorder; Depression; Social Stigma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy adolescents aged 13-18 years and adolescents aged 13-18 with current or remitted depression: The aim is to use a qualitative study design to investigate the spontaneous thoughts and feelings that young people express while viewing "ich bin alles" (English: "I am everything"; https://www.instagram.com/ich.bin.alles/) Instagram content.
  Purposive sampling is to be used for the study. In the case of this study, the targeted case selection refers to the age range (13-18 years) to be covered so that the study population contains participants from the entire age spectrum. In addition, the depression status (current or remitted depression or healthy) should be taken into account.
  Interventions: Behavioral: "ich bin alles" (English: "I am everything")

INTERVENTIONS:
Behavioral: "ich bin alles" (English: "I am everything") — The web-based information platform "ich bin alles" (www.ich-bin-alles.de) on depression and mental health in youth as well as its social media channels were developed by the Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy of the Ludwig-Maximilians-University Munich Hospital together with the Prof. Otto Beisheim Foundation. It is aimed at youth with depression, healthy youth, and their parents. The project focuses on education, prevention, low-threshold support, and destigmatisation through the transfer of evidence-based knowledge and hands-on supportive materials. Information material on Instagram is posted four times a week in the form of a post, a longer explanatory video and two reels (i.e., short videos with overlays of text and music; https://www.instagram.com/ich.bin.alles/). All content is evidence-based information created by the research team and is primarily based on the "ich bin alles" page.

SUMMARY:
Depression is a common mental disorder among adolescents, with increased rates during the COVID-19 pandemic. Despite its high burden, few young people seek professional help due to, among other things, low mental health literacy and fear of stigma. Since most adolescents often seek health information online and use social media daily, the "ich bin alles" (English: "I am everything"; www.ich-bin-alles.de) project was launched to provide accessible, age-appropriate information about depression via a website and social media channels (e.g., Instagram). This study aims to understand how participants perceive and evaluate the social media channel "ich bin alles" (English: "I am everything"; https://www.instagram.com/ich.bin.alles/).

DETAILED DESCRIPTION:
Depression is one of the most common mental disorders worldwide, with a prevalence of approx. 7.5% in youth. In connection with the COVID-19 pandemic, a meta-analysis found an increase in clinically relevant depressive symptoms to 25.2% in children and adolescents. At the same time, adolescents who experience mental health crises are reluctant to seek help and only 12% of adolescents with clinically relevant depressive symptoms seek professional treatment. The main barriers for young people to seek professional help include low knowledge of mental disorders/low mental health literacy and social factors such as the fear of stigmatization. Mental health literacy (MHL) is defined as "knowledge of how to prevent mental disorders, recognition of when a disorder is developing, knowledge of help-seeking options and treatment available, knowledge of effective self-help strategies for milder problems, and first aid skills to support others who are affected by mental health problems". It has been found that increased depression literacy can reduce depressive symptoms in adults and improve help-seeking for depression. Stigma in the context of mental health is a multidimensional concept that encompasses several domains. For many people living with mental illness, stigma is a significant contributor to a wide range of negative outcomes, including delayed help-seeking, hopelessness, diminished self-esteem, reduced quality of life and poorer clinical outcomes. Many of these negative effects have also been found in young people with mental health problems. Therefore, improving MHL and reducing the stigmatization of mental illness are two important starting points that can serve as targets for interventions. Improved MHL goes hand in hand with better knowledge about seeking help and less stigmatization of mental illness.

The vast majority of adolescents in western countries, such as the United States and Germany, have access to digital devices, such as smartphones. 97% of young people in the United States (13-17 years) state that they use social media and 45% say that they are online almost all the time. Along with this, young people are more likely to ask health questions, including mental health questions, online than through other channels. However, to date, few digital psychoeducational interventions for depression in adolescents have been developed and evaluated. In order to meet this need for action in a contemporary manner that attracts youth, the web-based project "ich bin alles" (English: "I am everything"; www.ich-bin-alles.de) was launched in September 2021 with an associated social media presence. The "ich bin alles" project provides comprehensive evidence-based and age-appropriate information on depression and mental health in youth via social media (such as Instagram). This strategy of providing information via social media is to be scientifically evaluated in this study.

The aim of this qualitative study is to evaluate the spontaneous thoughts and feelings that young people express while viewing "ich bin alles" Instagram content and to understand how the participants perceive and evaluate it. This will be investigated using the "Thinking Aloud Protocol"- method in 10-20 healthy adolescents and adolescents with current or remitted depression aged 13-18 years. The results of the study can help to gain insight into the perception and acceptance of the content.

ELIGIBILITY:
Inclusion Criteria:

* Ownership of an Instagram account
* Regular use of Instagram
* in group of adolescents with a current or remitted depression: ICD-10 diagnoses F32.0; F32.1; F32.2, F33.0, F33.1, F.33.2 based on "Diagnostisches Interview bei psychischen Störungen im Kindes- und Jugendalter (Diagnostic Interview for Mental Disorders in Childhood and Adolescence)"

Exclusion Criteria:

* Insufficient knowledge of German
* Following the "ich bin alles" (English: "I am everything") social media channels before participating in the study
* Knowing the "ich bin alles" (English: "I am everything") website before participating in the study
* in group of healthy adolescents: no ICD-10 diagnoses based on "Diagnostisches Interview bei psychischen Störungen im Kindes- und Jugendalter (Diagnostic Interview for Mental Disorders in Childhood and Adolescence)"

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 10-20 healthy adolescents and adolescents with current or remitted depression aged 13-18 years
  The study population will also be further described using the following questionnaires:
  1. Depression Literacy - Assessed with an adapted version of the German version of the Adolescent Depression Knowledge Questionnaire and the Depression Literacy Scale German (Time Frame: Start of appointment, before the Thinking Aloud Protocol)
  2. Stigma - Assessed with the German version of the Self Stigma of Depression Scale and an adapted Version of the Peer mental health stigmatization scale (Time Frame: Start of appointment, before the Thinking Aloud Protocol)
  3. Mental Health - Assessed with the Depression Screener for Teenagers and the Perceived Stress Scale (Time Frame: Start of appointment, before the Thinking Aloud Protocol)
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
spontaneous thoughts and feelings | during the 30 minutes in which the young people watch "ich bin alles" (English: "I am everything") content
  spontaneous thoughts and feelings that young people express while viewing "ich bin alles" Instagram content (English: "I am everything"; https://www.instagram.com/ich.bin.alles/)

SECONDARY OUTCOMES:
Acceptance | Day 1 (after the Thinking Aloud Protocol)
  questions (in form of a Semi-Structured Interview) designed by the investigators based on "the theoretical framework of acceptability"

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Schulte-Körne, Prof. Dr., Principal Investigator — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, LMU University Hospital
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, Hospital of the Ludwig-Maximilians-University (LMU) Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Consider briefly explaining why IPD will not or might not be shared. The data collected in this study include sensitive details about participants, such as various sociodemographic characteristics and information about mental health status. Publicly sharing the raw dataset could risk revealing individual identities, thereby violating ethical standards related to participant confidentiality. As a result, the raw data will not be publicly released. However, detailed descriptions of the methodology, materials used, and sample characteristics will be provided within the article and supplementary materials. The intervention is also publicly accessible in German on the "ich bin alles" - Instagram channel. Aggregated data and additional supporting materials may be shared upon request (contact: sara.kaubisch@med.uni-muenchen.de).

REFERENCES:
- See also: "ich bin alles" website — https://www.ich-bin-alles.de/
- See also: "ich bin alles" Instagram — https://www.instagram.com/ich.bin.alles/